CLINICAL TRIAL: NCT00655226
Title: Prevention of Depression in HIV/HCV Co-infected Substance Abuse Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low enrollment
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Thomas McGinn, MD, MPH, Mount Sinai School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO# 05-0961; R21DA021531 (NIH)
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Hepatitis C; Depressive Disorder, Major; Depressive Disorder; Depression; HIV Infections
Keywords: Cognitive Behavior Therapy; Interferon-alpha; Communicable Diseases; Liver Diseases; Depression; Hepatitis, Chronic; Interferons; Ribavirin; Hepatitis, Viral, Human; Infection; Hepatitis; Mood Disorders; Peginterferon alfa-2a; Hepatitis C; Interferon Alfa-2a; Interferon Alfa-2b; Depressive Disorder, Major; Depressive Disorder
MeSH Terms: conditions — Hepatitis C; Depressive Disorder, Major; Depressive Disorder; Depression; HIV Infections; Communicable Diseases; Liver Diseases; Hepatitis, Chronic; Hepatitis, Viral, Human; Infections; Hepatitis; Mood Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT skills based group sessions (Experimental): Cognitive Behavioral Therapy skills based group sessions
  Interventions: Behavioral: Cognitive Behavioral Therapy skills based group sessions
- Hepatitis C educational support groups (Active Comparator): Hepatitis C educational support groups
  Interventions: Behavioral: Hepatitis C educational support groups

INTERVENTIONS:
Behavioral: Hepatitis C educational support groups — Hepatitis C educational support groups
  Arms: Hepatitis C educational support groups
Behavioral: Cognitive Behavioral Therapy skills based group sessions — Eight CBT group sessions tailored for hepatitis C patients conducted by a clinical psychologist: 3 sessions conducted prior to IFN/ribavirin initiation, 1 session the day of IFN/ribavirin initiation, and 4 sessions during IFN/ribavirin treatment.
  Arms: CBT skills based group sessions

SUMMARY:
The purpose of this study is to determine whether cognitive behavioral therapy (CBT) is effective in the prevention of depression during interferon and ribavirin treatment for hepatitis C infection.

DETAILED DESCRIPTION:
The treatment for active hepatitis C in both HCV mono-infected and HCV/HIV co-infected patients is a long and difficult course, involving combination therapy of interferon and ribavirin for 6 to 12 months, a therapy with significant side effects. Up to 40% of patients being treated will develop depression due to the medication, which in turn leads to discontinuation of therapy and lost opportunities to prevent end stage liver disease. In fact, the presence of depression prior to interferon treatment often excludes patients from receiving interferon therapy, thereby denying them a potentially life-saving treatment. Non-pharmacological therapies such as cognitive behavioral therapy (CBT) have demonstrated efficacy in treating primary depression in numerous studies including in patients under going treatment with chronic medical illness. CBT is a well-established treatment modality and has been shown in several large randomized trials to be as effective, and in some cases more effective, than antidepressants. CBT has also shown efficacy in preventing the development of depression and other emotional disorders in high-risk populations. Offering CBT prior to and during treatment with interferon to non-depressed patients is a unique method that may reduce rates of depression and increase adherence to treatment without exposing patients to the risk of an additional medication.

ELIGIBILITY:
Inclusion Criteria:

1. >21 years
2. Speak and read English to 5th grade level of higher.
3. Eligible and ready to begin Peg-Interferon and Ribavirin (PEG-IFN/RBV) therapy for HCV at Mount Sinai's Primary Care practice or JMFC
4. HIV infected patients will need to have a CD4 count > 100 and have demonstrated compliance to retroviral therapy
5. Not majorly depressed upon entry to study.
6. Signed informed consent to participate in CBT study

Exclusion Criteria:

1. Majorly depressed (based on administration of the PHQ-9, score considered for Major Depressive Disorder).
2. Admit to actively abusing illicit drugs or alcohol
3. Medical contraindications to a standard course of interferon/ribavirin therapy (eg: severe anemia, uncontrolled congestive heart failure)
4. Less than one year of life expectancy
5. Current participation in CBT related psychotherapy
6. Participation in any psychotherapy beginning less than 6 months before CBT sessions begin.
7. Initiated anti-depressant medication less than 6 months before CBT sessions begin
8. Severe comorbid psychiatric disease including bipolar disorder, severe personality disorder, or psychotic disorder
9. Active suicidal ideation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Depression measured by PHQ-9 | study baseline, treatment visits (0, 2, 4, 8, 12, 18, 24, 30, 36, 42, and 48 weeks)
Depression measured by PHQ-9 | treatment visit 0 week
Depression measured by PHQ-9 | treatment visit 2 weeks
Depression measured by PHQ-9 | treatment visit 4 weeks
Depression measured by PHQ-9 | treatment visit 8 weeks
Depression measured by PHQ-9 | treatment visit 12 weeks
Depression measured by PHQ-9 | treatment visit 18 weeks
Depression measured by PHQ-9 | treatment visit 24 weeks
Depression measured by PHQ-9 | treatment visit 30 weeks
Depression measured by PHQ-9 | treatment visit 36 weeks
Depression measured by PHQ-9 | treatment visit 42 weeks
Depression measured by PHQ-9 | treatment visit 48 weeks

SECONDARY OUTCOMES:
Depressive symptoms (measured by Beck Depression Inventory-II) | study baseline, treatment visits (0, 2, 4, 8, 12, 18, 24, 30, 36, 42, and 48 weeks)
Depressive symptoms (measured by Beck Depression Inventory-II) | treatment visits 2 weeks
Depressive symptoms (measured by Beck Depression Inventory-II) | treatment visits 4 weeks
Depressive symptoms (measured by Beck Depression Inventory-II) | treatment visits 8 weeks
Depressive symptoms (measured by Beck Depression Inventory-II) | treatment visits 12 weeks
Depressive symptoms (measured by Beck Depression Inventory-II) | treatment visits 18 weeks
Depressive symptoms (measured by Beck Depression Inventory-II) | treatment visits 24 weeks
Depressive symptoms (measured by Beck Depression Inventory-II) | treatment visits 30 weeks
Depressive symptoms (measured by Beck Depression Inventory-II) | treatment visits 36 weeks
Depressive symptoms (measured by Beck Depression Inventory-II) | treatment visits 42 weeks
Depressive symptoms (measured by Beck Depression Inventory-II) | treatment visits 48 weeks
medication adherence | study baseline
medication adherence | treatment visits 0 week
medication adherence | treatment visit 2 weeks
medication adherence | treatment visit 4 weeks
medication adherence | treatment visit 8 weeks
medication adherence | treatment visit 12 weeks
medication adherence | treatment visit 18 weeks
medication adherence | treatment visit 24 weeks
medication adherence | treatment visit 30 weeks
medication adherence | treatment visit 36 weeks
medication adherence | treatment visit 42 weeks
medication adherence | treatment visit 48 weeks
hepatitis C treatment completion | study baseline
hepatitis C treatment completion | treatment visit 0 week
hepatitis C treatment completion | treatment visit 2 weeks
hepatitis C treatment completion | treatment visit 4 weeks
hepatitis C treatment completion | treatment visit 8 weeks
hepatitis C treatment completion | treatment visit 12 weeks
hepatitis C treatment completion | treatment visit 18 weeks
hepatitis C treatment completion | treatment visit 24 weeks
hepatitis C treatment completion | treatment visit 30 weeks
hepatitis C treatment completion | treatment visit 36 weeks
hepatitis C treatment completion | treatment visit 42 weeks
hepatitis C treatment completion | treatment visit 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G McGinn, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States